CLINICAL TRIAL: NCT01438905
Title: Effect of Joint Mobilization on Muscle Activation and Function in Individuals With Chronic Ankle Instability
Brief Title: Effect of Joint Mobilization in the Treatment of Chronic Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Collaborators: Nebraska Foundation for Physical Therapy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 11-16058
Record Dates: First submitted 2011-09-14; First posted 2011-09-22 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Ankle Sprain
Keywords: Ankle Sprain; Chronic Ankle Instability; Ankle Mobilization; Talocrural Joint Mobilization; Cortical Muscle Activation; Spinal Muscle Activation
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Parameters will be identical to the lower intensity (Small amplitude oscillation mobilization; Grade IV) talocrural mobilization. No force, other than light hand contact will be applied by the therapist.
- Lower intensity mobilization (Experimental): The subject will be in a seated position and the therapist will stabilize the distal tibia with one hand and make contact the anterior talus with the opposite hand. Three 60-second anterior to posterior joint mobilizations of the talus (small amplitude at end range; Grade IV) will be applied by the therapist with one minute rest in between sets.
  Interventions: Other: Small amplitude (Grade IV) mobilization
- Higher intensity mobilization (Experimental): The subject will be in a seated position and the therapist will grasp the dorsum of the foot with their fingers. The ankle will be dorsiflexed until the restrictive barrier is reached. A small amplitude, quick thrust at end of range (High velocity, low amplitude; Grade V mobilization/manipulation) will be applied. If joint cavitation is not felt or heard by the therapist or subject the technique will be repeated one additional time.
  Interventions: Other: High velocity, low amplitude (Grade V) mobilization

INTERVENTIONS:
Other: Small amplitude (Grade IV) mobilization — The subject will be in a seated position and the therapist will stabilize the distal tibia with one hand and make contact the anterior talus with the opposite hand. Three 60-second anterior to posterior joint mobilizations of the talus (small amplitude at end range; Grade IV) will be applied by the therapist with one minute rest in between sets.
  Arms: Lower intensity mobilization
Other: High velocity, low amplitude (Grade V) mobilization — The subject will be in a seated position and the therapist will grasp the dorsum of the foot with their fingers. The ankle will be dorsiflexed until the restrictive barrier is reached. A small amplitude, quick thrust at end of range (High velocity, low amplitude; Grade V mobilization/manipulation) will be applied. If joint cavitation is not felt or heard by the therapist or subject the technique will be repeated one additional time.
  Other Names: Manipulation; Grade V mobilization; High velocity, low amplitude thrust
  Arms: Higher intensity mobilization

SUMMARY:
The purpose of this study is to examine the effects of a gentle pressure movement performed at the ankle by a physical therapist on muscle function and ankle motion in individuals who frequently twist (sprain) their ankle.

DETAILED DESCRIPTION:
Novel rehabilitation methods, that specifically target decreased muscle activation due to joint pathology prior to strength training, have elicited greater improvements in muscle function and self-reported disability compared to traditional therapies. Preliminary evidence suggests ankle joint mobilization can improve contributions of spinal influences on ankle muscle activation in individuals with ankle joint pathology, but there is a considerable gap in understanding cortical contributions to muscle activation following joint injury. It is unknown how joint mobilization concurrently affects cortical and spinal neural motor pathways, as well as clinical measures of patient function. The overall aim of this grant is to determine the immediate effects of talocrural joint mobilization on cortical and spinal muscle activation of the fibularis longus (peroneus) and soleus muscles in individuals with chronic ankle instability (CAI). The secondary aims of this study will examine changes in ankle dorsiflexion range of motion (ROM) and dynamic balance. This innovate approach will provide the necessary scientific knowledge regarding the potential mechanism and efficacy of joint mobilization.

ELIGIBILITY:
Inclusion Criteria:

* Age 16-45 years
* History of one or more ankle sprains
* Scoring at least an 85% on the Foot and Ankle Ability Measure (FAAM) Sport or at least 3 on the Modified Ankle Instability Instrument (AII).
* At least 5° ankle dorsiflexion asymmetry compared to the contralateral limb OR ankle dorsiflexion ROM less than 21°

Exclusion Criteria:

* Lower extremity injury or surgery within the past 6 months (including lateral ankle sprain)
* Diagnosed ankle osteoarthritis
* History of ankle surgery that involves intra-articular fixation
* Medical conditions which would be contraindications to mobilization/manipulation and/or transcranial magnetic stimulation, including cardiac pacemaker, metal implants in the head, current pregnancy, neurological disorders, recent use of stimulants or medications known to lower seizure threshold, and personal or family history of seizures

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-09; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Changes in Muscle activation | Baseline and immediately after each manual therapy intervention; 1 week study
  To determine cortical and spinal changes in muscle activation of the fibularis longus and soleus following one of three intervention protocols. Changes in cortical and spinal muscle activation will be measured by examining resting motor threshold via Transcranial Magnetic Stimulation and the H-reflex technique, respectively.
  The investigators hypothesize that the higher intensity talocrural joint mobilization will result in a greater increase in cortical and spinal activation of the fibularis longus and soleus muscles than the lower intensity talocrural joint mobilization.
Changes in Ankle dorsiflexion ROM | Baseline and immediately after each manual therapy intervention; 1 week study
  To determine the changes in ankle dorsiflexion ROM following one of two talocrural joint mobilization techniques (higher or lower intensity) or control intervention in individuals with CAI. Changes in ankle dorsiflexion ROM will be quantified using a weight bearing lunge.
  The investigators hypothesize that the higher intensity (Grade V) talocrural joint mobilization will result in a greater improvement in ankle dorsiflexion ROM than the lower intensity (Grade IV) talocrural joint mobilization and the control intervention will result in no change in ROM.
Changes in Dynamic Balance | Baseline and immediately after each manual therapy intervention; 1 week study
  To determine the acute changes in balance following one of two talocrural joint mobilization techniques or control intervention in individuals with CAI. Changes in balance will be quantified using the anterior, posteromedial, and posterolateral components of the Star Excursion Balance Test.
  The investigators hypothesize that the higher intensity talocrural joint mobilization will result in greater improvements in reach distance in all three SEBT directions compared to the lower intensity talocrural joint mobilization.

CONTACTS AND LOCATIONS:
Overall Officials: Terry L Grindstaff, PhD, PT, ATC, Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States

REFERENCES:
- [Derived] Grindstaff TL, Dolan N, Morton SK. Ankle dorsiflexion range of motion influences Lateral Step Down Test scores in individuals with chronic ankle instability. Phys Ther Sport. 2017 Jan;23:75-81. doi: 10.1016/j.ptsp.2016.07.008. Epub 2016 Jul 29. PMID 27662790